CLINICAL TRIAL: NCT04441359
Title: Effects of the Supplementation With Oligosaccharides on the Prevention of Infections in Infants
Brief Title: Long-term Safety and Efficacy of Prebiotic Enriched Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: Laboratorios Ordesa (Industry); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Study protocol June 2008 final
Record Dates: First submitted 2020-06-10; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Infection; Microbial Colonization; Healthy
MeSH Terms: conditions — Infections; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplemented formula (Experimental): Standard formula supplemented with prebiotic inulin-type fructans
  Interventions: Other: Supplemented formula
- standard formula (Placebo Comparator): Standard Formula not supplemented with prebiotic inulin-type fructans
  Interventions: Other: Standard formula

INTERVENTIONS:
Other: Supplemented formula — standard infant formula supplemented with 8 g/L prebiotic inulin-type fructans
  Arms: supplemented formula
Other: Standard formula — standard infant formula not supplemented with prebiotic inulin-type fructans
  Arms: standard formula

SUMMARY:
The primary objective of the present study was to evaluate the effects of long-term supplementation of an infant formula supplemented with prebiotic inulin-type oligosaccharides on immunological-health related outcomes.

DETAILED DESCRIPTION:
The study primarily aimed to evaluate the effects of long-term supplementation of an infant formula with a mixture of short and long chain inulin-type oligosaccharides on immunological-health related outcomes, as well as on gastrointestinal function and well-being in infants during the first year of life. Effects on infant growth, tolerance and on the composition of fecal microbiota were further objectives of this study. The study was conducted as a multicenter, randomised, double-blind, placebo-controlled study in healthy term infants. The two groups of the study are product group (standard infant formula supplemented with inulin-type fructans) and control group (non-supplemented standard infant formula).

ELIGIBILITY:
Inclusion Criteria:

* Healthy babies born between 37 - 42 weeks of gestation and with weight appropriate for gestational age (between percentiles 3 and 97)
* Healthy babies aged between 0 - 4 months of age
* Babies exclusively fed with an infant formula on enrolment into the study

Exclusion Criteria:

* The presence of an infection at the moment of the recruitment or 1 week before recruitment
* The presence of important pathologies (intestinal, cardiopathy, mental retardation, etc.)
* Any other diseases related to the immune system (primary immunodeficiency)
* Parents not able to comply with the study follow up (according to physician criteria)

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2010-10-31 (Actual); Study Completion 2010-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of infections during first year of life | until infant reaches age of 1 year
  measured through presence of fever, and number and duration of infectious episodes

SECONDARY OUTCOMES:
Stool frequency | until infant reaches age of 1 year
  Number of depositions per day assessed by parenteral reporting (parent's diary collected during first week of each study month throughout all study period)
Stool consistency | until infant reaches age of 1 year
  Assessed via 1-3 scale with pictograms (1=hard, 2=soft/formed, 3=liquid/semi-liquid), by parenteral reporting (parent's diary collected during first week of each study month throughout all study period)
Digestive tolerance | until infant reaches age of 1 year
  Number of vomiting and regurgitation episodes per day and presence of excessive flatulence and infantile colic, assessed by parenteral reporting (parent's diary collected during first week of each study month throughout all study period)
Growth | until infant reaches age of 1 year
  Calculation of z-scores of weight-for-age and length-for-age according to the World Health Organisation (WHO) standards using WHO software (WHO Antro software).
Body weight | until infant reaches age of 1 year
  Assessment of weight (kg) of the nude infant via calibrated electronic scales at all study visits.
Body height | until infant reaches age of 1 year
  Assessment of height (cm) in supine position by using a standard measuring board at all study visits.
Head circumference | until infant reaches age of 1 year
  Assessment of head circumference (cm) using a non-extendable insertion tape at all study visits.
Sleeping habits | until infant reaches age of 1 year
  Assessment of total hours slept and total hours of nocturnal sleeping per day (min), by parenteral reporting (parent's diary collected during first week of each study month throughout all study period).
Crying episodes | until infant reaches age of 1 year
  Assessment of crying episodes (min), by parenteral reporting (parent's diary collected during first week of each study month throughout all study period).
Effect on fecal microbiota composition | until infant reaches age of 1 year
  Quantification of dominant bacterial groups
Effect on development of allergy | until infant reaches age of 1 year
  Presence of clinical symptoms compatible with food allergies, atopic dermatitis, exanthema
Effect on immunology markers in feces | until infant reaches age of 1 year
  secretory immunoglobulin A, calprotectin level

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - ZNA Koningin Paola Kinderziekenhuis, Antwerp
  - Universitair Ziekenhuis, Brussels
- Spain (6):
  - CAP Llefià, Barcelona
  - Hospital de Nens, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital San Cecilio, Granada
  - Equipo Pediátrico San Francisco, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodriguez-Palmero, M.; Campoy, C.; Urraca, O.; Alonso, J.; Maldonado, J.; Varea, V.; Palencia, J.; Veereman-Wauters, G.; Neumer, F.; Rivero, M.; Vandenplas, Y. Effects of long-term supplementation with a mixture of short and long chain inulin-type oligosaccharides (2013), Annals of Nutrition and Metabolism, suppl. 1, (63), 1-1960.